CLINICAL TRIAL: NCT03360916
Title: Impact of Statin Therapy on Adaptations to Aerobic Exercise
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00140791; R01AR071263 (NIH)
Record Dates: First submitted 2017-11-20; First posted 2017-12-04 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases
Keywords: high cholesterol; exercise; statins
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia; Motor Activity | interventions — Atorvastatin; Tablets; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo & Exercise Group (Placebo Comparator): Participants randomized to this group will undergo placebo treatment and an aerobic exercise program.
  Interventions: Drug: Placebo; Behavioral: Exercise Program
- Low Statin & Exercise Group (Experimental): Participants randomized to this group will undergo low statin treatment (Lipitor 20Mg Tablet) and an aerobic exercise program.
  Interventions: Drug: Lipitor 20Mg Tablet; Behavioral: Exercise Program
- High Statin & Exercise Group (Experimental): Participants randomized to this group will undergo high statin treatment (Lipitor 80Mg Tablet) and an aerobic exercise program.
  Interventions: Drug: Lipitor 80Mg Tablet; Behavioral: Exercise Program

INTERVENTIONS:
Drug: Lipitor 20Mg Tablet — One tablet by mouth every day for 12 weeks.
  Other Names: Atorvastatin
  Arms: Low Statin & Exercise Group
Drug: Lipitor 80Mg Tablet — One tablet by mouth every day for 12 weeks.
  Other Names: Atorvastatin
  Arms: High Statin & Exercise Group
Drug: Placebo — One matching placebo tablet by mouth every day for 12 weeks.
  Arms: Placebo & Exercise Group
Behavioral: Exercise Program — Exercise program of brisk walking and/or slow jogging on a treadmill for 90 minutes of exercise spread over 3 days during week 1, 150 minutes of exercise spread over 5 days during week 2, 225 minutes of exercise over 5 days during week 3 and for the rest of the study.

SUMMARY:
The purpose of this study is to determine how different doses of a statin affect muscle health and exercise.

DETAILED DESCRIPTION:
High cholesterol and cardiovascular disease (CVD) is currently prevented and treated with statin therapy. Statin use can cause muscle weakness, fatigue and/or pain, and these symptoms can increase with dose and duration of statin use. Statins may also change the ability to exercise.

This study is testing how different doses of a statin, Lipitor, affect muscle health and exercise. The doses that will be used in this study (20 mg/day or 80 mg/day) are typical for treating high cholesterol.

This study is expected to last about 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 25-43 kg^m2
* Sedentary (less than 150 min of physical activity/week during last 6 months)
* Weight stable (no more than 5% change in body weight the previous 3 months)

  * >5% risk for a cardiovascular event in the next 10 years according to the 2013 American College of Cardiology/American Heart Association risk calculator and/or 2 out of 5 metabolic syndrome risk factors(Triglycerides ≥ 150 mg/dL; HDL ≤ 40 mg/dL; Glucose ≥ 100mg/dL; Waist Circumference ≥ 102cm for males, 88cm for females; Blood pressure: ≥ 130mmHg systolic and/or 85mmHg diastolic or being treated for hypertension).
* Stable doses of medications for 90 days
* Willing to stop all Nonsteroidal Antiinflammatory Drugs (NSAIDs) and aspirin for 7 days prior to muscle biopsy

Exclusion Criteria:

* Smoking
* Use of statins in the last 6 months
* Use of other medications or supplements that affect lipid profiles or body weight in the last 6 months (e.g., fibric acids, bile acid sequestrants, nicotinic acids, fish oil)
* Diagnosis of chronic diseases including CVD, diabetes, other metabolic diseases (e.g., thyroid), cancer, HIV, or acquired immunodeficiency syndrome
* History of abnormal bleeding problems
* Currently taking (within the last 10 days) anti-platelet medication (Plavix), Warfarin, and other anti-coagulants (eliquis, pradaxa, and xarelto) medications
* >2 fold upper normal limit (UNL) for alanine aminotransferase (ALT) or creatinine
* Women who are pregnant or breastfeeding
* Individuals with polymorphisms known to be associated with susceptibility for statin induced myopathies (tested at screening)
* Currently enrolled in another research study

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Thyfault, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 52 participants that were officially enrolled were randomized
Groups:
- Placebo: Participants receiving matching placebo oral tablet.
  Placebo Oral Tablet: Matching placebo pill.
- Low Dose Statin: Participants will receive Lipitor 20Mg Tablet to take daily.
  Lipitor 20Mg Tablet: 20 mg/day pills.
- High Dose Statin: Participants will receive Lipitor 80Mg Tablet to take daily.
  Lipitor 80Mg Tablet: 80 mg/day pills.
Period: Overall Study
Arm/Group | Placebo | Low Dose Statin | High Dose Statin
Started | 16 | 17 | 19
Completed | 14 | 13 | 16
Not Completed | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Low Dose Statin: Participants receiving Lipitor 20Mg Tablet to take daily.
  Lipitor 20Mg Tablet: 20 mg/day pills.
- High Dose Statin: Participants receiving Lipitor 80Mg Tablet to take daily.
  Lipitor 80Mg Tablet: 80 mg/day pills.
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose Statin | High Dose Statin | Total
Number analyzed (Participants) | 16 | 17 | 19 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.13 (8.29) | 51.28 (9.04) | 50.85 (7.96) | 50.78 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 15 | 40
  Male | 4 | 4 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 4 | 12
  White | 10 | 13 | 14 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 19 | 52
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 200.19 (31.63) | 220.33 (38.54) | 204.90 (32.24) | 208.65 (34.72)
Weight [Mean (Standard Deviation); unit: kg] | 94.74 (16.15) | 103.42 (20.06) | 95.83 (14.33) | 98.10 (17.08)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.68 (4.58) | 35.43 (5.14) | 34.55 (4.84) | 34.88 (4.79)
Relative Peak VO2 Max [Mean (Standard Deviation); unit: mL/kg/min] | 25.29 (6.21) | 21.30 (6.27) | 22.74 (5.74) | 22.97 (6.15)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Mitochondrial Respiratory Function
Time Frame: Value at 3 months minus value at baseline
Measure: Mean (Standard Deviation); unit: pmols/s/mg
Arm/Group | Placebo | Low Dose Statin | High Dose Statin
Number analyzed (Participants) | 11 | 10 | 14
pmols/s/mg | 2.29 (125.59) | -11.24 (130.12) | 44.88 (105.19)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.9530, t-test, 2 sided; This is within group 3 month change; Mean Difference (Net) = 2.29, Standard Deviation 125.59
Statistical Analysis 2: Comparison: Low Dose Statin; Test type: Superiority; p = 0.7908, t-test, 2 sided; This is within group 3 month change; Mean Difference (Net) = -11.24, Standard Deviation 130.12
Statistical Analysis 3: Comparison: High Dose Statin; Test type: Superiority; p = 0.1344, t-test, 2 sided; This is within group 3 month change; Mean Difference (Net) = 44.88, Standard Deviation 105.19

2. Secondary Outcome: Change in VO2 Max
Time Frame: Value at 12 months minus value at baseline
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Placebo | Low Dose Statin | High Dose Statin
Number analyzed (Participants) | 14 | 13 | 16
L/min | 0.22 (0.18) | 0.23 (0.21) | 0.21 (0.23)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.0005, t-test, 2 sided; This is within group 3 month change; Mean Difference (Net) = 0.22, Standard Deviation 0.18
Statistical Analysis 2: Comparison: Low Dose Statin; Test type: Superiority; p = 0.0021, t-test, 2 sided; This is within group 3 month change; Mean Difference (Net) = 0.23, Standard Deviation 0.21
Statistical Analysis 3: Comparison: High Dose Statin; Test type: Superiority; p = 0.0025, t-test, 2 sided; This is within group 3 month change; Mean Difference (Net) = 0.21, Standard Deviation 0.23

ADVERSE EVENTS:
Time Frame: Participants were contacted weekly by phone or email and prompted to disclose any adverse events. Additional adverse events could be reported if participant contacted study team outside of the usual weekly check in. Adverse events were monitored until symptoms subsided or adverse event ended or until the end of the 12 month intervention period.
Arm/Group | Placebo | Low Dose Statin | High Dose Statin
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 3/16 | 5/17 | 8/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Low Dose Statin (N=17) | High Dose Statin (N=19)
Muscle or Joint Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 7 (7)
Restless Legs (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory Illness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The COVID-19 epidemic started in the middle of the trial forcing us to stop recruitment for four months. Furthermore, the continuation of the pandemic slowed recruitment for the rest of the trial and significantly impacted n size. There was also a national dextrose shortage following a hurricane in Puerto Rico. As a result many of the IVGTT were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT03360916/Prot_SAP_000.pdf